CLINICAL TRIAL: NCT03208387
Title: Biological Substrates of Impaired Neurocognitive Functioning: Understanding the Late Effects of Surviving a Pediatric Brain Tumor
Brief Title: Understanding the Late Effects of Surviving a Pediatric Brain Tumor
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Columbia University (Other); University of Washington (Other); University of Texas (Other); Rutgers University (Other)
Responsible Party: Sponsor
Other Study IDs: 17-338
Record Dates: First submitted 2017-06-29; First posted 2017-07-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Brain Tumor; Pediatric Brain Tumor; Pediatric Cancer
Keywords: 17-338; Cognitive function; Behavioral function
MeSH Terms: conditions — Brain Neoplasms; Neoplasms | interventions — Diffusion Tensor Imaging; Wechsler Scales; Memory and Learning Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children Medulloblastoma Survivors: Participants previously treated for M0 non-disseminated medulloblastoma with cranio-spinal irradiation plus a boost to the posterior fossa
  Interventions: Diagnostic Test: Diffusion tensor imaging (DTI); Diagnostic Test: Resting state functional connectivity MRI (rs-fcMRI); Behavioral: Wechsler Intelligence Scale for Children - 5th edition (WISC-V); Behavioral: California Verbal Learning Test (CVLT-C); Behavioral: Beery Test of Visual Motor Integration 6th edition; Behavioral: Grooved Pegboard; Behavioral: PedsQL Multidimensional Fatigue Scale; Diagnostic Test: MRI
- Children Astrocytoma Survivors: Participants previously treated for a low grade cerebellar astrocytoma, with surgery only and neither chemotherapy nor cranial irradiation.
  Interventions: Diagnostic Test: Diffusion tensor imaging (DTI); Diagnostic Test: Resting state functional connectivity MRI (rs-fcMRI); Behavioral: Wechsler Intelligence Scale for Children - 5th edition (WISC-V); Behavioral: California Verbal Learning Test (CVLT-C); Behavioral: Beery Test of Visual Motor Integration 6th edition; Behavioral: Grooved Pegboard; Behavioral: PedsQL Multidimensional Fatigue Scale; Diagnostic Test: MRI
- Age-Matched Healthy Children Controls
  Interventions: Behavioral: Wechsler Intelligence Scale for Children - 5th edition (WISC-V); Behavioral: California Verbal Learning Test (CVLT-C); Behavioral: Beery Test of Visual Motor Integration 6th edition; Behavioral: Grooved Pegboard; Behavioral: PedsQL Multidimensional Fatigue Scale; Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: Diffusion tensor imaging (DTI) — DTI quantifies the degree to which water diffuses in different directions through a given brain region. The use of DTI as an in vivo index of the integrity of white matter has been applied to many disease states using several proprietary and open-source software programs (e.g. FSL 5.0). DTI tractography, employed via toolboxes such as Probtrackx within the FSL 5.0, allows the identification of white matter tracts connecting cortical and subcortical regions of interest. Furthermore, structural connectivity as measured with DTI does not duplicate functional connectivity as measure with rs-fcMRI, but rather provides complimentary perspectives.
  Groups: Children Astrocytoma Survivors; Children Medulloblastoma Survivors
Diagnostic Test: Resting state functional connectivity MRI (rs-fcMRI) — rs-fcMRI is a relatively new neuroimaging technique that has been applied to studying multiple clinical populations including ADHD, schizophrenia, major depressive disorder, and other neurological disorders. The approach exploits measurement of changes in brain blood oxygenation (BOLD) as is employed in task based functional MRI (measuring changes in focal cortical vascular oxygenation when engaged in a defined task, e.g. motor movement). Neuroimaging data will be collected as soon as possible (can be the same day), for up to 6 weeks.
  Groups: Children Astrocytoma Survivors; Children Medulloblastoma Survivors
Behavioral: Wechsler Intelligence Scale for Children - 5th edition (WISC-V) — Will gather IQ data and is the gold standard for IQ assessment for those between the ages of 6:0 and 16:11 years.
  Other Names: WISC-V
Behavioral: California Verbal Learning Test (CVLT-C) — Validated measure of verbal learning and memory for those between the ages of 5:0 and 16:11.
  Other Names: CVLT-C
Behavioral: Beery Test of Visual Motor Integration 6th edition — Measure designed to assess visual-motor functioning of subjects between the ages of 2-99 years old by copying designs using paper and pencil.
Behavioral: Grooved Pegboard — This is a standard assessment of fine motor functioning and dexterity by asking the subject to place metal pegs into holes on a board.
Behavioral: PedsQL Multidimensional Fatigue Scale — Designed to measure fatigue in pediatric patients (ages 5-17 years) and is comprised of the General Fatigue Scale (6 items), Sleep/Rest Fatigue Scale (6 items) and Cognitive Fatigue Scale (6 items).
Diagnostic Test: MRI — Images will be acquired on a 3.0 Tesla MRI scanner at each of the four study sites. At MSK, resting state fMRI data will be obtained using a 3T GE scanner with an 8-channel head coil (Discovery 750w DV25)

SUMMARY:
The goal of this study is to learn about the cognitive and behavioral functioning of children being treated for cancer.

ELIGIBILITY:
Inclusion Criteria:

Children Treated for Posterior Fossa Tumors:

* As per medical record or clinical report, successfully completed all medical treatment for either an M0 posterior fossa medulloblastoma without dissemination or posterior fossa low-grade astrocytoma without relapse or evidence of residual disease.
* For medulloblastoma survivors only: Previously treated with gross total resection (GTR), craniospinal irradiation with conformal posterior fossa boost radiotherapy (CSI + Boost) and chemotherapy
* For low grade astrocytoma survivors only: Previously treated with gross total resection ONLY (no chemotherapy or radiotherapy).
* As per medical record or clinician report, between 1-10 years post completion of their medical treatment for their posterior fossa brain tumor.
* Subject is between the ages of 6 through 16 years at time of consent.
* As per medical record or parent report, subject is able to tolerate an MRI without sedation.

Healthy Control Participants:

* No major medical illness, as determined by medical interview by study physician.
* As per parent report, subject is between the ages of 6 through 16 years at time of consent.
* As per parent report, subject is able to tolerate an MRI without sedation.

Exclusion Criteria:

All Participants:

* Full Scale IQ as documented to be below a standard score of <70 based upon the study IQ assessment completed after consent.
* As per self or parent report, completed any portion of the neuropsychological battery used in this study within the last year.
* MRI contraindications (e.g., implanted ferromagnetic devices, claustrophobia) as per radiology clinical operating procedures.
* As per self or parent report or medical record, currently taking medications that have CNS effects (i.e., antidepressants, neuroleptics, anti-seizure medications, drugs that affect blood pressure or heart rate, alpha-agonists, adrenergic blockers, lithium, sedating antihistamines, and some medications for the treatment of asthma).
* As per self or parent report, non-fluency in English language as demonstrated by current educational placement in a non-English-speaking classroom setting.

Ages: 6 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Participants will be recruited at MSK and three participating sites (Columbia University, University of Washington and University of Texas Southwestern).
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibilty which is the number of eligible survivors consented per month | 2 years
  The study is a pilot study to collect information on feasibility broadly defined. The feasibility indicators are primarily descriptive variables, including a careful monitoring of accrual rate (how many eligible survivors consented per month).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Sands, PsyD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org